CLINICAL TRIAL: NCT02217683
Title: Pulmonary Hemodynamic Effects of Stored Red Blood Cell Transfusion in Post-Operative Cardiac Surgical Patients: Influence of Breathing Nitric Oxide. A Randomized Controlled Trial in the Cardiac-Intensive Care Unit.
Brief Title: Use of Inhaled Nitric Oxide to Prevent Pulmonary Hypertension Associated to Stored Blood Transfusion
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This trial never started due to lack of funding.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Staff anesthesiologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BloodiNO
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension, Pulmonary; Hemolysis
Keywords: Catheterization, Swan-Ganz; Cardiac Surgical Procedures; Blood Transfusion; Nitric Oxide
MeSH Terms: conditions — Hypertension, Pulmonary; Hemolysis | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Young blood transfusion (No Intervention): The first group of patients (n=30) will be randomized to receive leukoreduced blood transfusion stored for less than 10 days
- Old blood transfusion (No Intervention): This randomized group of patients (n=30) will receive leukoreduced blood transfusion stored for more than 30 days
- Old blood transfusion and Nitric Oxide (Active Comparator): This randomized group of patients (n=30) will receive leukoreduced blood transfusion stored for more than 30 days while breathing nitric oxide (80 part per million) and oxygen
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Nitric oxide at 80 part per million will be administrated by inhalation for approximately 1 hour during the blood transfusion
  Arms: Old blood transfusion and Nitric Oxide

SUMMARY:
The objective of this study is to assess if prolonged storage time of a packed red blood cell unit may cause pulmonary vasoconstriction after transfusion, in a susceptible population such as cardiac surgery patients. The investigators will also evaluate the potential reversal effect of Inhaled Nitric Oxide on pulmonary vasoconstriction induced by stored blood transfusions.

DETAILED DESCRIPTION:
Patients will be randomized into one of the three groups:

I. Blood transfusion stored for less than 10 days II. Blood transfusion stored for more than 30 days III. Blood transfusion stored for more than 30 days days plus inhalation of Nitric Oxide at 80 part per million for an hour during blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Elective cardiac or aortic surgery
3. One or more blood transfusions scheduled for clinical reasons
4. Presence of an arterial catheter and pulmonary arterial catheter

Exclusion Criteria:

1. Emergent cardiac surgery.
2. Patients requiring irradiated or washed blood transfusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vascular resistance index | During and after blood transfusion- average time of observation 6 hours
  Parameters to calculate pulmonary vascular resistance index will be measured during and after blood transfusion for about 6 hours. The following parameters will be recorded: height, weight, systemic pressure, pulmonary pressure, wedge pressure, central venous pressure, cardiac output) of each subjects will be recorded.

SECONDARY OUTCOMES:
Hemolysis | During and after blood transfusion- average time of observation 6 hours
  Hemolytic markers will be measured such as: haptoglobin, plasma free hemoglobin, hemopexin, and iron metabolites.
Nitric oxide metabolites | During and after blood transfusion- average time of observation 6 hours
  Plasma nitric oxide consumption, plasma and red blood cell levels of circulating nitrate, nitrite, nitric will be measured
Inflammation | During and after blood transfusion- average time of observation 6 hours
  Inflammation will be assessed by changes of the plasma concentration of cytokines, such as IL-6, IL-8, IL-10, IL-12, TNF, IFN-γ

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Berra L, Pinciroli R, Stowell CP, Wang L, Yu B, Fernandez BO, Feelisch M, Mietto C, Hod EA, Chipman D, Scherrer-Crosbie M, Bloch KD, Zapol WM. Autologous transfusion of stored red blood cells increases pulmonary artery pressure. Am J Respir Crit Care Med. 2014 Oct 1;190(7):800-7. doi: 10.1164/rccm.201405-0850OC. PMID 25162920